CLINICAL TRIAL: NCT06796842
Title: Effects of Ballistic vs Plyometric Training on Performance of Badminton Players
Acronym: EBVPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nadia Ishtiaq
Record Dates: First submitted 2025-01-10; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sports Physical Therapy
Keywords: badminton; performance; ballistic; plyometrics
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballistic group (Other): Ballistic training program was set for 6 weeks. Each week consisting of 5 exercises with sets of 3 and repetitions of 10,15 and 20 times, recovery time and training intensity differed each week.
  Interventions: Other: Ballistic Exercises
- Plyometric Group (Experimental): Plyometric training program was set for 6 weeks. With four exercises in 1st week. Five in 2nd and 3rd weeks, six exercises in 4th and seven exercises in last two weeks. Each exercise consisted of 3 sets with 10, 15 and 20 repetitions in each. Recovery time and training intensity differed each week.
  Interventions: Other: Plyometric exercises

INTERVENTIONS:
Other: Ballistic Exercises — Ballistic training program was set for 6 weeks. Each week consisting of 5 exercises with sets of 3 and repetitions of 10,15 and 20 times, recovery time and training intensity differed each week.
  Arms: Ballistic group
Other: Plyometric exercises — Plyometric training program was set for 6 weeks. With four exercises in 1st week. Five in 2nd and 3rd weeks, six exercises in 4th and seven exercises in last two weeks. Each exercise consisted of 3 sets with 10, 15 and 20 repetitions in each. Recovery time and training intensity differed each week.
  Arms: Plyometric Group

SUMMARY:
Ballistic and plyometric training are both frequently utilized to enhance physical performance in a variety of sporting activities that require the ability to jump, sprint, and change direction. both are designed to improve explosive power, but they differ in their approaches and focus. Although many studies highlight the significance of both plyometric and ballistic exercises in enhancing athletic performance in badminton players no direct comparison has been made between the two.

In this study we compared the effectiveness of Ballistic exercises versus Plyometric exercises on performance in Badminton players, which is going to help us to select the best possible training program for badminton athletes

DETAILED DESCRIPTION:
Ballistic and plyometric training are both frequently utilized to enhance physical performance in a variety of sporting activities that require the ability to jump, sprint, and change direction. both are designed to improve explosive power, but they differ in their approaches and focus. Although many studies highlight the significance of both plyometric and ballistic exercises in enhancing athletic performance in badminton players no direct comparison has been made between the two.

In this study we compared the effectiveness of Ballistic exercises versus Plyometric exercises on performance in Badminton players, which is going to help us to select the best possible training program for badminton athletes

ELIGIBILITY:
Inclusion Criteria

* Active Badminton player.
* Age between 20-28 years.
* Male Badminton players

Exclusion Criteria

* Athletes with injuries, trauma, pathology, any neurological or psychological complications.
* Athletes with Metabolic diseases.
* Age above 28 years or less than 20.
* Other than male Players.

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Push up test | six weeks
  The Test demanded that the test subject lie face down on the floor with their elbows pointing backward down their side, their hands beneath their shoulders, and their fingers pointing forward. The individual's body weight rested on their hands and toes after pushing themselves to full arm extension; The up position was this. Then, maintaining a straight body, the person lowered himself until the entire body, from the chest to the thighs, made contact with the ground. Then the participants returned to the up position after being pulled up to full arm extension. One push-up test was made up of these up and down steps. from enrollment to the end of treatment up to six weeks
Closed kinetic chain upper extremity stability test | six weeks
  On a tiled floor, athletic tape strips were positioned 36 inches apart and parallel to one another. The test began with one hand in the push-up position on each piece of tape. From the beginning, the patients were told to reach across their body with one hand and touch the piece of tape underneath the other hand. The hand was put back in the beginning position after touching the tape line. The patient then used the other hand to make the same motion. The testing lasted 15 seconds in total. from enrollment to the end of treatment up to six weeks
Seated medicine ball throw test | six weeks
  Each athlete started the test by holding the 2 kg medicine ball with both hands, resting it firmly against their chest. The task was to throw the ball forward as far as possible using a chest press motion, a movement that primarily engages the chest, shoulders, and arms in an effort to achieve maximum distance. from enrollment to the end of treatment up to six weeks
Unilateral single arm shot put test | six weeks
  To evaluate upper body strength and power, a 3-kilogram medicine ball was used. On the floor, athletes sat with their feet flat, knees bent at a 90-degree angle, and backs against the wall on the floor for stability. They were positioned next to a doorway to allow unrestricted arm movement on the test side. The participants were instructed to hold the medicine ball at shoulder height and push it forward-rather than throwing it-using an explosive chest press motion to propel it as far as possible. from enrollment to the end of treatment up to six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nadia Ishtiaq, MS, Study Director — Riphah International University
Locations (1):
- Liaqat Bagh Stadium Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This article focuses on the current concepts of plyometric exercises and their application in sports therapy. The goal of the article is to explore the principles, benefits, and methods of plyometric training in the context of athletic performance — https://pmc.ncbi.nlm.nih.gov/articles/PMC4637913/
- See also: This study explores the impact of a specific plyometric training program, known as "Ballistic Six," on the performance of medium-pace bowlers in cricket. The focus is on Asian Indian cricket bowlers who typically require explosive strength and speed — https://www.researchgate.net/publication/326625710_The_Effect_of_'Ballistic_Six'_Plyometric_Training_on_Performance_of_Medium_Pace_Asian_Indian_Cricket_Bowlers
- See also: This study explores the impact of ballistic exercises (exercises involving explosive movements) over an eight-week training period, specifically focusing on their effects on muscle power. — https://pubmed.ncbi.nlm.nih.gov/18815571/
- See also: likely focusing on the differences in performance outcomes and how each type of exercise influences the mechanical aspects of the bench press movement, such as force production, velocity, and power output. — https://pubmed.ncbi.nlm.nih.gov/28225524/